CLINICAL TRIAL: NCT02779972
Title: Age Related Changes in Cardiac Physiology as a Predictor of Exercise Tolerance
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director. Research & Development, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-16-UC-0090-16-TLV-CTIL
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Aging; Exercise Tolerance
Keywords: Cardiac Physiology; Physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 60's decade: 60's decade Echo stress test
  Interventions: Other: Echo stress test
- 70's decade: 70's decade Echo stress test
  Interventions: Other: Echo stress test
- 80's decade: 80's decade Echo stress test
  Interventions: Other: Echo stress test

INTERVENTIONS:
Other: Echo stress test — Echo stress test

SUMMARY:
Aging is associated with numerous changes and adaptations in the cardiovascular system. Vascular and ventricular wall thickness increase, whereas arterial compliance, endothelial function, and ventricular contractility decline. The decline in cardiac function with advancing age is typically seen in parallel to reduced physical activity, and it has been proposed that lifelong exercise training might attenuate the effects of aging on the heart.

The cardiovascular system undergoes several age-related changes. For most healthy older individuals, the heart generally functions well under resting conditions. Structural and physiological changes tend to result in diminished exercise tolerance. However, increasingly it has been shown that even some of these changes are more a result of a sedentary lifestyle than an age-related phenomenon. Most elderly people tend to become less physically active. It is difficult to separate changes intrinsic to the aging process from those arising as a result of a sedentary lifestyle.

DETAILED DESCRIPTION:
Previous large studies have concluded that resting LV diastolic and systolic function decline with age. The cardiovascular system undergoes several age-related changes. For most healthy older individuals, the heart generally functions well under resting conditions. Structural and physiological changes tend to result in diminished exercise tolerance. However, increasingly it has been shown that even some of these changes are more a result of a sedentary lifestyle than an age-related phenomenon. Most elderly people tend to become less physically active. It is difficult to separate changes intrinsic to the aging process from those arising as a result of a sedentary lifestyle. Studies of aging and physical activity usually compare older athletes with sedentary ones, in which physical activity was not found to attenuate the impact on the aging heart. Thus, the investigators set of to find the difference between hearts of elderly who are physically fit as measured with METS to those who are not. And try and understand the basis of this difference.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 65 with preserved systolic function and stress echo on a treadmill between 1 Jan 2012 until 31 Dec 2015 in the facility.

Exclusion Criteria:

* Missing complete information used for data collection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients above 65 with preserved systolic function and stress echo on a treadmill between 1 Jan 2012 until 31 Dec 2015 in our facility
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-04 (Actual)

PRIMARY OUTCOMES:
Cardiac output at maximal stress test | 45 minutes
  mean cardiac output in liter per minute for each age group

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Chorin, MD, Principal Investigator — 972-3-6947520
Locations (1):
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No